CLINICAL TRIAL: NCT00485888
Title: Changes in the Vasodilatory Response to Methyl-nicotinate in Response to S-citalopram Treatment in Social Phobia Patients
Brief Title: Flushing in Social Anxiety Disorder on Cipralex
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: START Clinic for Mood and Anxiety Disorders (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Principal Investigator, Dr. Martin A. Katzman, Principal Investigator, START Clinic for Mood and Anxiety Disorders
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LuCipMNSP
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2008-10

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social | interventions — Dexetimide; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Cipralex
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cipralex — 10-20mg; one per day
  Other Names: Escitalopram
  Arms: 1
Drug: Placebo — Matched to Cipralex
  Arms: 2

SUMMARY:
To add to our understanding of the relationship between blushing, symptom severity and potential mechanisms that underlie blushing in patients with SP, we propose comparing SP patients' vascular responses to topical m-N pre and post treatment with S-citalopram or placebo.

S-citalopram (an SSRI) has been widely used in the treatment of mood and anxiety disorders as it has shown efficacy in these patients (Lepola et al., 2003; Stahl et al., 2003; Burke et al., 2002; Davidson et al., 2002; Wade et al., 2002). In comparison to placebo, S-citalopram has been shown to be effective and well tolerated in those with short and long term SP (Lader et al 2004; Montgomery et al., 2003; Kasper et al., 2002). As indicated, responses to the blushing exposure will be assessed prior to and following treatment with S-citalopram or placebo and at one month following the intervention.

Levels of prostaglandin will be compared between groups and will also be correlated with symptom severity in the clinical groups. Effective psychological interventions that reduced the fear of blushing in individuals with social phobia did not lead to a reduction in actual blushing during a social test (Mulkens et al., 2001). As such, it is expected that the patients' perception of amount of blushing will change following treatment. In addition, we are undertaking an investigation as to whether nican topical administration will change following treatment to match the pattern seen in healthy controls.

The objectives are to evaluate the efficacy of S-citalopram 10 to 20 mg once daily (QD) in the treatment of social phobia and to determine if treatment outcome is related changes in intensity of the vasodilatory response to 10 mM topical m-N. This is a randomized, double-blind flexible-dose study evaluating the efficacy, safety and tolerability of S-citalopram 10 to 20 mg and placebo in outpatient subjects diagnosed with SP. At the screening visit those who are eligible will enter a randomized trial with S-citalopram 10 to 20 mg and placebo. The study will begin with a single week of S-citalopram 10 mg. Subsequently, capsules will be administered in a flexible dose fashion and patients will be followed up weekly (biweekly after week 6) and at the clinician's discretion. After the first week the patients' dosage will be increased up to a maximum of 20 mg daily. This dose will remain fixed after 8 weeks of treatment until week 16.

DETAILED DESCRIPTION:
Objectives

The objectives are to evaluate the efficacy of S-citalopram 10 to 20 mg once daily (QD) in the treatment of social phobia and to determine if treatment outcome is related changes in intensity of the vasodilatory response to 10 mM topical m-N.

Study Population

Out-patients (n = 36) with a primary diagnosis of Social Phobia using DSM-IV criteria (300.02), with or without other comorbid secondary illnesses, who meet all other inclusion/exclusion criteria are eligible to enter the study. We have chosen to assign 36 completed subjects as the number of desired completers. Given a drop out rate of 20%, 44 subjects will be enrolled in the study.

Study Design

This is a randomized, double-blind flexible-dose study evaluating the efficacy, safety and tolerability of S-citalopram 10 to 20 mg and placebo in outpatient subjects diagnosed with SP. At the screening visit those who are eligible will enter a randomized trial with S-citalopram 10 to 20 mg and placebo. The study will begin with a single week of S-citalopram 10mg. Subsequently, capsules will be administered in a flexible dose fashion and patients will be followed up weekly (biweekly after week 6) and at the clinicians discretion. After the first week the patients' dosage will be increased up to a maximum of 20 mg daily. This dose will remain fixed after 8 weeks of treatment until week 16.

Voluntary discontinuation by a subject

Subjects are free to discontinue their participation in the study at any time, without prejudice to further treatment. Subjects who discontinue from the study should always be asked about the reason(s) for their discontinuation and the presence of any adverse events. If possible, they should be seen and assessed by an investigator. Adverse events will be followed up.

Safety Evaluation:

Once treatment phase is initiated and 30 days following the conclusion of the trial, subjects will be questioned on any adverse events related to administration of S-citalopram. At the final visit, 30 days after the conclusion of the trial, patients will be given a full physical examination. Adverse experiences will be documented in response to a non-leading question such as, "Have you felt different in any way since starting the new treatment or since the last visit?" In addition, all adverse experiences observed by the investigator or volunteered spontaneously by the patient will be recorded. Any serious adverse events (SAE) will be reported to H. Lundbeck A/S contact person within 24 hours of becoming aware of them.

Serious Adverse Events meets at least one of the following indicators:

1. Death
2. Life threatening
3. In patient hospitalization
4. Persistent or significant disability/ incapacity
5. Congenital anomaly/birth defect
6. Judged medically important

Efficacy Evaluation:

Primary efficacy parameter

The primary objective is as follows:

In individuals with SP, changes in intensity of the vasodilatory response to 10 mM topical m-N will be measured in association with symptomatic improvement following treatment with S-citalopram 10 to 20 mg. The end point of the study period is Week 16.

Secondary efficacy parameters

The secondary objectives are as follows and the end point of the study period is Week 16:

1. Mean change from baseline on the Liebowitz Social Anxiety Scale (LSAS); Hamilton Anxiety Scale (HAM-A), Social Phobia Inventory (SPIN); Beck Anxiety Inventory (BAI); Social Phobia Scale (SPS) at final visit; and the Social Interaction Anxiety Scale (SIAS)
2. Mean change from baseline on fear of blushing scales: Blushing, Trembling, and Sweating Questionnaire (BTS-Q) and Propensity Scale (BPS).
3. Decreased levels of prostaglandin D2 will be observed in association with the findings of decreased m-N -induced flushing in the SP population. Any significant differences in levels of prostaglandin D2 and its metabolite between the three groups (treatment group and the controls) will disappear with symptom improvement in the SP group.
4. Potential changes in peripheral serotonin synthesis from tryptophan will be altered such that changes in levels of plasma serotonin will be correlated with outcome and flushing response in SP subject who received treatment.
5. Mean change from baseline on the Sheehan Disability Scale (work, social life and family life domains), Euroquol (quality of life) and the Medical Outcomes Study Short-Form-36 (SF-36), ), Penn State Worry Questionnaire (PSWQ)

Trial Design:

This is a randomized, double-blind flexible-dose study evaluating the efficacy, safety and tolerability of S-citalopram 10 to 20 mg and placebo in outpatient subjects diagnosed with SP.

After providing written informed consent at the screening visit, the patient will undergo all tests indicated to determine suitability for the study. Patients meeting all inclusion/exclusion criteria will then be assigned to receive S-citalopram (N = 18) or placebo (N = 18). The initial dose of S-citalopram will be 10mg. After week one, patients will be managed on a dose of 10mg daily to a maximum of 20mg. The dose may be adjusted for the first 8 weeks and then kept stable for duration of the rest of the study. Patients will be seen weekly from week one to 6 and biweekly until week 16, and if necessary, telephone contact will be initiated by the Investigator or study coordinator between visits to assess the patient's response to therapy.

Procedure for Assessing Blushing/Vasodilation:

Prior to application of each m-N patch, a 5 mm diameter circle of relatively hairless, unblemished skin will be masked off with hypoallergenic medical tape. This area will be found on both the subjects' inner forearm and face (center of cheekbone - below the outside corner of the eye). Initially, a five-minute baseline laser Doppler measurement will be taken. Subsequently, the 10 mM m-N patch will be applied over the skin area on the forearm or face for one minute and then removed. This is followed by a 20-minute period during which blood flow will be measured continuously over both the face and arm.

Vasodilatation will be measured by using a Moor Instruments moorLAB laser Doppler spectroscope adjusted to measure changes in cutaneous blood flow. The Laser Doppler flow meter takes real time measurements of local tissue blood flow by reflecting light off a moving object such as a red blood cell. Each measurement will then be assigned an arbitrary unit (Flux) which is a parameter based on the summed intensity of reflections recorded by the instrument (Moor Instruments Limited, 1998). Flux will be sampled 40 times per second and transferred to a personal computer for analysis.

Subsequently, blood flow (flux) data will be averaged into 30-second bins and analyses will be undertaken using non-linear curve fitting using the software program Prism (Graphpad software). The flux at any time t [F(t)] will be fitted to a curve with parameters F(0), the baseline flux, F, the maximal plateau change in flux, µ, the maximal rate of change, and L, the lag time between applying the test patch and vasodilatation occurring (Equation 1). Runs which do not produce a significant reaction (this being defined as at least one block of 5 consecutive 30 second time periods being significantly (Student's t-test; P < 0.05) above baseline blood flow) will be assigned a F value of zero; the µ and L parameters can not be calculated in these circumstances).

Approximate half maximal dose (EC50) values will be calculated using non-linear curve fitting to a standard sigmoidal dose response curve using the median F values derived from each dose of m-N.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for this trial are patients who meet all of the following criteria:

  1. The patient has provided signed informed consent.
  2. Outpatients aged 18-65 (extremes included).
  3. Patients with a primary diagnosis of Social Phobia according to DSM IV (300.23) criteria (diagnosis to be made using the Mini International Neuropsychiatric Interview (MINI)).
  4. On the basis of a physical examination, medical history and basic laboratory screening, the patient is, in the investigators opinion, in a suitable condition.
  5. Willing and able to attend study appointments in the correct time windows.

Exclusion Criteria:

* Patients meeting one or more of the following criteria cannot be selected for inclusion:

  1. Any other axis I diagnosis that was a primary disorder in the previous six months.
  2. Continuation or commencement of formal psychotherapy.
  3. Alcohol or drug abuse as defined in the DSM IV within the last six months.
  4. Mania or hypomania as defined in the DSM IV.
  5. Current use of or commencement of antidepressant and anxiolytic medications.
  6. Patients, who have been on an antidepressant or other anxiolytic prior to the study, will have discontinued it more than two weeks prior to entry into the study. Those who have been on fluoxetine, will have been off of it for at least 5 weeks
  7. Patients who have been on an herbal or alternative treatment judged to be potentially anxiolytic or with psychobiological activity, will have terminated usage of the agent more than two weeks prior to entering the study.
  8. Previous reaction to Niacin administration
  9. Use of a non-steroidal anti-inflammatory
  10. Any psychotic disorder.
  11. Eating disorders as defined in the DSM IV.
  12. Mental retardation or other cognitive disorder.
  13. Clinical interpretation of apparent suicide risk.
  14. Laboratory values at screening or in medical history that may be considered through clinical interpretation to be significant.
  15. Diseases which could, through clinical interpretation, interfere with the assessments of safety, tolerability and efficacy.
  16. Serious illness: Liver or renal insufficiency, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurological, infectious, neoplastic or metabolic disturbance.
  17. The patient is, in the opinion of the investigator, unlikely to be able to comply with the clinical trial protocol, or is unsuitable for any other reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Changes in intensity of the vasodilatory response to 10 mM topical m-N over 16 weeks. | 20 weeks

SECONDARY OUTCOMES:
Mean change from baseline on the LSAS, HAM-A, SPIN,BAI, SPS, SIAS, BTS-Q, BPS,Sheehan Disability Scale, Euroquol SF-36, PSWQ | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin A Katzman, MD, Principal Investigator — START Clinic for the Mood and Anxiety Disorders
Locations (1):
- START Clinic for the Mood and Anxiety Disorders, Toronto, Ontario, Canada